CLINICAL TRIAL: NCT02267759
Title: A Comparison of McGrath Videolaryngoscopy and Macintosh Laryngoscopy for Routine Nasotracheal Intubation
Brief Title: McGrath Videolaryngoscopy for Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AJIRB-DEV-DE1-14-312
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- McGrath (Experimental): Nasotracheal intubation was performed with McGrath videolaryngoscopy
  Interventions: Device: Macintosh laryngoscopy
- Macintosh (Active Comparator): Nasotracheal intubation was performed with Macintosh direct laryngoscopy
  Interventions: Device: McGrath videolaryngoscopy

INTERVENTIONS:
Device: McGrath videolaryngoscopy — After the softened nasotracheal tube was inserted into the nares until its tip passed through the posterior nares, McGrath videolaryngoscope was introduced into the mouth and the nasotracheal tube was advanced.
  Arms: Macintosh
Device: Macintosh laryngoscopy — After the softened nasotracheal tube was inserted into the nares until its tip passed through the posterior nares, Macintosh laryngoscope was introduced into the mouth and the nasotracheal tube was advanced.
  Arms: McGrath

SUMMARY:
McGrath videolaryngoscopy avoids the use of Magill forceps for nasotracheal intubation, thereby reducing intubation time and complications, especially in patients with a difficult airway. This study was performed to investigate whether McGrath videolaryngoscopy is superior to Macintosh laryngoscopy for routine nasotracheal intubation in expected normal airways, as judged by the time to intubation and ease of intubation.

ELIGIBILITY:
Inclusion Criteria:

* patients for dental or maxillofacial surgery requiring nasotracheal intubation

Exclusion Criteria:

* known difficult airway
* required rapid sequence induction
* history of bleeding
* cervical spine injury

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
time to intubation | 4 min after anesthetic induction
  time the nasotracheal tube was inserted into nares until endtidal CO2 was detected

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea